CLINICAL TRIAL: NCT06899178
Title: A Phase 2, Double Blind, Randomized, Placebo-controlled Crossover Trial to Evaluate the Efficacy and Safety of Atomoxetine in Adults With Melanocortin Obesity Syndrome
Brief Title: Atomoxetine in Melanocortin Obesity Syndrome
Acronym: MCOS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Joan Han, Professor of Pediatrics, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 24-0669
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Melanocortin Obesity Syndrome; MCOS
Keywords: Obesity; BDNF; MC4R; Atomoxetine; Energy balance; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, crossover study of atomoxetine. The treatment periods will last 16 weeks, separated by a 2-week washout period. Atomoxetine immediate release is approved for treatment of ADHD in children and adults. Enrollment will be based on age groups in batches, beginning with 10 adults, to optimize the protocol and monitor safety/efficacy before treating younger patients. If safety and efficacy are acceptable, the pediatric cohort will be enrolled. The intervention length of 16 weeks per arm was chosen to allow for 4 weeks of dose titration and 12 weeks exposure to target dose. The FDA effectiveness threshold for anti-obesity medication is 5% weight loss after 12 weeks. The half-life of atomoxetine is approximately 5 hours. A two-week washout period will allow for elimination of study drug while minimizing participant burden from frequent study visits.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo then Atomoxetine (Placebo Comparator): Participants receive placebo for 16 weeks (4 weeks titration + 12 weeks at target dose), followed by washout period, then atomoxetine for 16 weeks (4 weeks titration + 12 weeks at target dose).
  Interventions: Drug: Atomoxetine; Drug: Placebo
- Atomoxetine then Placebo (Active Comparator): Participants receive atomoxetine for 16 weeks (4 weeks titration + 12 weeks at target dose), followed by washout period, then placebo for 16 weeks (4 weeks titration + 12 weeks at target dose).
  Interventions: Drug: Atomoxetine; Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Initial dose 40 mg, day 7 dose 60 mg, day 14 dose 80 mg, day 21 dose 100 mg (target dose)
Drug: Placebo — Matching placebo oral capsule

SUMMARY:
This is a phase 2 randomized placebo-controlled crossover trial to determine the safety and efficacy of atomoxetine for treating obesity caused by loss-of-function variants in the melanocortin-4 receptor (MC4R), the most common cause of genetic obesity disorders. Atomoxetine was selected for this pilot trial because it has been shown to increase brain-derived neurotrophic factor (BDNF) within the central nervous system and in peripheral circulation. Targeting BDNF is a specific strategy for treating MC4R abnormalities because BDNF functions as a downstream mediator of MC4R signaling.

DETAILED DESCRIPTION:
Targeted therapies for the treatment of monogenetic obesity are essential because typical lifestyle interventions and standard anti-obesity medications are largely ineffective as they do not correct the specific genetic defect causing abnormal energy balance. The leptin pathway is the key regulator of body weight through control of appetite and energy expenditure. In particular, the severe insatiable hunger experienced by patients with leptin pathway disorders leads not only to extreme obesity, but the unrelenting drive to seek food also causes substantial distress for patients and caregivers. While therapies have been developed for treating genetic disorders affecting the proximal portion of the leptin pathway (LEP, LEPR, POMC, PCSK1, and BBS1-22), there are no treatments for loss-of-function LOF) variants of the melanocortin-4 receptor gene (MC4R), which cause melanocortin obesity syndrome (MCOS). In various population and cohort studies, 1-6% of patients with severe, early onset obesity are found to have MC4R LOF variants, making MCOS the most common cause of genetic obesity. Brain-derived neurotrophic factor (BDNF) is a downstream mediator of MC4R signaling and, therefore, may serve as a specific target for MCOS treatment. The researchers propose repurposing a well-understood and commercially available attention-deficit hyperactive disorder (ADHD) medication, atomoxetine (FDA-approved for the treatment of ADHD in persons ages 6 years and older), for the treatment of MCOS because of animal and human studies show that this drug induces endogenous BDNF levels. Atomoxetine could potentially increase hypothalamic BDNF levels, leading to weight loss through improved anorectic signaling downstream of the abnormally functioning MC4R. A phase 2 randomized, placebo-controlled crossover trial in 20 patients with MCOS will be conducted to test this hypothesis. The study will begin in adult patients and if safety and efficacy are shown, then pediatric patients age ≥ 6 years will be studied. The primary outcome measure will be change in BMI (expressed as the percentage of the 95th percentile BMI for age/sex). Additional measures will include percent body fat and visceral fat area by bioelectrical impedance analysis, resting energy expenditure by indirect calorimetry, dietary intake by food frequency questionnaire and 24-hour recall, hyperphagia score, hunger level, satiety level, hemoglobin A1c, lipid panel, liver function tests, blood pressure, heart rate, and ADHD symptoms. Serum and plasma BDNF and genetic variants in atomoxetine metabolism enzymes will be assessed and correlated with weight changes. This pilot clinical trial will provide valuable data on the safety and efficacy of atomoxetine for treating MCOS, and the data will be used to guide the design of a future phase 3, multicenter, randomized clinical trial.

ELIGIBILITY:
Inclusion criteria:

* Age 6 years and above
* Documented MC4R variant classified as pathogenic, likely pathogenic, or variant of uncertain significance per ACMG criteria. If testing was done in a research lab, it will be confirmed by a CLIA-approved lab prior to randomization.
* Obesity defined as BMI ≥30 kg/m2 in adults or ≥95th percentile for age and sex in children

Exclusion criteria:

* Use of atomoxetine, viloxazine (another selective norepinephrine-reuptake inhibitor), methylphenidate, amphetamine, dextroamphetamine, lisdexamfetamine, phentermine, or any other stimulant medication in the past 30 days. If on other ADHD medications, such as guanfacine and clonidine, must be on a stable dose for >3 months.
* Weight loss >5% in the past 3 months.
* Initiation of new weight loss program, including diet or medications. If on weight loss medications, must be on a stable dose for >3 months.
* Inability to swallow capsules.
* History of hypersensitivity to atomoxetine.
* Narrow angle glaucoma.
* History of pheochromocytoma.
* Uncontrolled Stage 2 hypertension (≥95th percentile + 12 mmHg or >140/90, whichever is lower) at screening. If on antihypertensive medication, must be on stable dose for >3 months.
* Hepatic insufficiency including cirrhosis and acute hepatitis (AST or ALT >3x upper limit of normal)
* Uncontrolled asthma requiring albuterol more than once weekly over the past 3 months
* History of a cardiac arrhythmia (not including bradycardia)
* Current use of monoamine oxidase inhibitors
* Pregnancy or intention to become pregnant during the next year
* History of Major Depressive Disorder in the past 2 years, lifetime history of suicide attempt, history of any suicidal behavior in the past month, history of other severe psychiatric disorders (e.g. schizophrenia, bipolar disorder)
* PHQ-9 score is ≥15 or suicidal ideation of type 4 or 5 (C-SSR) in the past month
* Unable to comply with study procedures in the opinion of the investigator

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 16 weeks
  BMI will be calculated as kg/sq m. The sex appropriate CDC growth chart will be used to calculate BMI as a percent of the 95th percentile (BMI95). For patients >20 years, the 20-year-old percentiles will be used.

SECONDARY OUTCOMES:
Resting Energy Expenditure (REE) | 16 weeks
  Resting energy expenditure (REE) will be measured by indirect calorimetry after a minimum 1 hour of rest in the Clinical Research Center. Oxygen consumption and carbon dioxide production will be measured. The first 5-10 minutes of data will be discarded to allow participants to adjust to the metabolic cart.
Healthy Eating Index (HEI) | 16 weeks
  The VioScreen assessment provides a Healthy Eating Index (HEI) score to measure the quality of a person's diet. The HEI score ranges from 0 to 100, with higher scores indicating better eating habits.
Hyperphagia Questionnaire (HQ) | 16 weeks
  Hyperphagia will be assessed with the Hyperphagia Questionnaire (HQ)
  This is a 13-item questionnaire with each question answered on a 5-point scale. Two of the questions are qualitative.
  Full range is scored from 11 to 55. Higher score indicates greater hyperphagia.
Hunger and Satiety Score | 16 weeks
  Full range scored from 0 to 10 with higher score indicating greater hunger/satiety.
Fasting Glucose Level | At week 0, week 16 and week 32.
  A blood sugar test measures the amount of a sugar called glucose in a sample of blood.
  Fasting laboratory studies will be obtained at week 0, week 16 and week 32.
Alanine Transaminase (ALT) Level | At week 0, week 16 and week 32.
  The alanine transaminase (ALT) blood test measures the level of the enzyme ALT in the blood. ALT is an enzyme found in a high level in the liver. An enzyme is a protein that causes a specific chemical change in the body.
  Fasting laboratory studies will be obtained at week 0, week 16 and week 32.
Fasting Insulin Level | At week 0, week 16 and week 32.
  The insulin level in blood. Insulin is a hormone produced by beta cells in the pancreas.
  Fasting laboratory studies will be obtained at week 0, week 16 and week 32.
Hemoglobin A1c | At week 0, week 16 and week 32.
  A1C is a lab test that shows the average level of blood sugar (glucose) over the previous 3 months. It shows how well blood sugar is controlled to help prevent complications from diabetes.
  Fasting laboratory studies will be obtained at week 0, week 16 and week 32.
Lipid Panel - Fasting LDL, HDL, Triglycerides | At week 0, week 16 and week 32.
  A lipid profile is a blood test to measure different types of lipids:
  High-density lipoprotein cholesterol (HDL [good] cholesterol): HDL helps remove LDL from your blood.
  Low-density lipoprotein cholesterol (LDL [bad] cholesterol): LDL can build up in your blood vessels and increase your heart disease risk.
  Triglycerides: Your body makes some triglycerides. Triglycerides also come from the food you eat. Extra calories are turned into triglycerides and stored in fat cells for later use.
  Fasting laboratory studies will be obtained at week 0, week 16 and week 32.
High Sensitivity C-Reactive Protein | At week 0, week 16 and week 32.
  C-reactive protein (CRP) is produced by the liver. The level of CRP rises when there is inflammation in the body. It is one of a group of proteins, called acute phase reactants that go up in response to inflammation. The levels of acute phase reactants increase in response to certain inflammatory proteins called cytokines. These proteins are produced by white blood cells during inflammation.
  The CRP test is a general test to check for inflammation in the body. It is not a specific test. A high-sensitivity C-reactive protein (hs-CRP) is a more A more sensitive CRP test
  Fasting laboratory studies will be obtained at week 0, week 16 and week 32.
The ASEBA Brief Problem Monitor | 16 weeks
  The ASEBA Brief Problem Monitor (BPM) is a quick assessment tool designed to monitor and track a child's behavioral and emotional problems over time, particularly focusing on internalizing, externalizing, and attention issues.
  Range is 0 to 99.9th percentile
Adult ADHD Self-Report Scale (ASRS-v1.1) Symptom Checklist. | 16 weeks
  This is an 18-item self-report questionnaire designed for individuals to assess their own symptoms of Attention Deficit Hyperactivity Disorder (ADHD) focusing on daily experiences related to attention, impulsivity, and hyperactivity. Total scale is scored 0-72 with higher score indicating more predictive of an ADHD diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Joan C Han, MD, Principal Investigator — Mount Sinai Kravis Children's Hospital; Ashley H Shoemaker, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Mount Sinai Hospital, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be included in the URL field below).
URL: https://dataverse.org/